CLINICAL TRIAL: NCT03056495
Title: Multicenter, Open-label Phase Ib Dose-escalation and Dose-confirmational Study for the Tolerability and Safety of N-hydroxy-N'-Phenyl-octanediamide (Vorinostat) in Patients With Mild Alzheimer's Disease
Brief Title: Clinical Trial to Determine Tolerable Dosis of Vorinostat in Patients With Mild Alzheimer Disease
Acronym: VostatAD01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Hospital, Bonn (Other); University of Göttingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VostatAD01; 2014-005311-17 (EudraCT Number)
Record Dates: First submitted 2016-12-27; First posted 2017-02-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Investigational drug (Experimental): N-hydroxy-N'-phenyl-octanediamide (Vorinostat) capsules once a day, three weeks of treatment; dose escalation with different dosages per cohort; One cohort of three subjects
  Interventions: Drug: N-hydroxy-N'-phenyl-octanediamide (Vorinostat)

INTERVENTIONS:
Drug: N-hydroxy-N'-phenyl-octanediamide (Vorinostat) — N-hydroxy-N'-phenyl-octanediamide capsules once a day, three weeks of treatment; dose escalation with different dosages per cohort; One cohort of three subjects
  Other Names: Vorinostat

SUMMARY:
This Clinical Trial is an open, non-randomized Phase Ib study to determine the maximal tolerable dose (MTD) of Vorinostat in Alzheimer disease (AD) patients between (including) 55 and 90 years with mild symptoms. The MTD in this study is defined as the dose that leads to maximum toxicity with Common Toxicity Criteria (CTC) grade 1 symptoms.The safety and tolerability of Vorinostat in this group of study participants should be tested.

DETAILED DESCRIPTION:
The MTD of Vorinostat in the treatment of Alzheimer's patients is to be determined by using an open, non-randomized, multicentric dose-finding study with adaptive design. This Clinical Trial will take place in 2 parts.

The first part will be performed as a dose escalation part in cohorts of three subjects. Possible dosages will be: one, two, three or four capsules (100 mg per capsule) once per day. The first cohort receives a dose of 100 mg per day. After the treatment, a Vorinostat-free follow-up phase will take place. For the following cohorts, dose increases, a repetition of the previous dose or a dose reduction are possible.

After the dose escalation with a determination of the MTD, a dosage confirmation is carried out with additional subjects. The subjects are given a dose of Vorinostat of MTD over 4 weeks followed by a Vorinostat-free follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate in the study
* verified capacity to consent by a doctor not involved in the study
* mild Alzheimer's disease (NINCDS / ADRDA criteria and Mini-Mental State Examination (MMSE) 22-27)
* age (including) from 55 to 90 years
* subjects must be able to meet the requirements described in the study protocol
* outpatient living
* Informant lives with subject in the same household
* Rosen modified Hachinski ischemia score ≤4
* concerning only female patients: postmenopausal
* concerning only male patients: commitment to use a suitable contraceptive
* cerebral imaging study (CT or cMRI), which is consistent with a diagnosis of probable Alzheimer's disease (not older than 3 years)

Exclusion Criteria:

* other neurological and psychiatric diseases explaining cognitive deficits better than an AD diagnosis
* conspicuous MRI / CCT scan explaining the cognitive deficits better than an AD diagnosis
* severe physical, neurological or psychiatric disorders that interfere with the participation in the study
* history of malignant tumors except non- metastasizing basal cell carcinoma of the skin
* history of seizures
* dysphagia leading to the inability to swallow capsules
* untreated severe acute infections with clinical symptoms such as respiratory infections, pneumonia, bronchitis, acute diarrhea, influenza, untreated urinary tract infections
* in the family history, unexplained sudden cases of heart failure before the age of 50 years
* long QT syndrome in the family history
* evidence of QTc prolongation ≥480 ms at screening (Fridericia adjusted QT interval), of arrhythmias especially of severe uncontrolled ventricular arrhythmias or atrial fibrillation in ECG
* not sufficiently treated angina
* heart failure (NYHA III, IV)
* myocardial infarction
* known infection with HBV, HCV and / or HIV
* occurrence of venous thrombosis or embolism
* therapy with antidepressants begun in the last 12 weeks or dose modification of a pre-existing therapy with antidepressants
* antidiabetic treatment begun in the last 12 weeks or dose modification of pre-existing antidiabetic treatment
* long-term use of anti-inflammatory drugs except acetylsalicylic acid for cardiovascular prophylaxis
* current treatment or treatment within the past 12 weeks with HDAC inhibitors (eg valproate)
* taking medication that may increase the dose-dependent side effects myelosuppression or QTc interval prolongation.

These include, but are not limited to:

* Class Ia antiarrhythmic agents such as quinidine, procainamide, disopyramide
* Class III antiarrhythmic drugs such as amiodarone, sotalol, ibutilide
* Class Ic antiarrhythmics such as flecainide, propafenone
* penicillamine
* opioids such as methadone and pyrazolone derivatives such as metamizole and Propyphenazone
* doxorubicin, epirubicin
* macrolides and their analogues such as erythromycin, clarithromycin
* telithromycin
* oxazolidinones such as linezolid
* quinolones such as moxifloxacin, levofloxacin
* fluoxetine, maprotiline
* tricyclic and tetracyclic antidepressants
* chlorpromazine, pimozide, haloperidol, droperidol, ziprasidone and clozapine
* antiemetics
* azole like ketoconazole, fluconazole, voriconazole
* aminocholine such as primaquine
* pentamidine such as quinine, chloroquine
* diaminopyrimidine such as pyrimethamine
* salbutamol and formoterol methotrexate
* azathioprine, cyclosporine Interferon gamma 1b
* alemtuzumab, basiliximab, efalizumab, natalizumab
* sunitinib, nilotinib, lapatinib
* mitoxantrone, Hydroxycarbamide, mercaptopurine
* taking of prescription and non-prescription drugs for cognitive enhancement (except cholinesterase inhibitors and memantine at a stable dose for at least 3 months before baseline)
* therapy with anticoagulants except acetylsalicylic acid
* HbA1c in screening more than 10% above the upper limit of normal
* magnesium, sodium, calcium and potassium levels outside the normal range (at screening and baseline)
* existing anemia with Hb <11 (at screening and baseline)
* existing thrombocytopenia; platelet ≤150.000 / ul, leukocytes ≤ 3.000 / ul, neutrophils absolutely ≤ 1.500 / ul (at screening and baseline)
* prothrombin or INR ≥ 1.5 above the laboratory limit of normal; PTT ≥ 1.5 x above the laboratory limit of normal (at screening and baseline)
* clinically relevant renal and / or hepatic impairment at screening and baseline (total bilirubin ≥ 1.5 x above the upper limit of the norm and / or GPT, AST ≥ 4x above the upper limit of the norm and / or creatinine ≥ 1.5x above the upper limit of the norm and / or creatinine clearance <60 ml / min)
* hematuria> 15 RBCs / mL at screening and baseline
* proteinuria at screening and baseline except in asymptomatic urinary tract infections
* participating in other clinical and therapeutic trials within the last 12 weeks

relevant only for dose confirmation:

* subjects with existing contraindications for performing an MRI if no MRI available from the period of 6 months prior to screening
* cardiac pacemaker
* metal objects in the body, which exclude a 1.5 or 3 T MRI
* claustrophobia

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum-tolerated dose (MTD) in elderly subjects during dose escalation | 12 months
  A MTD is defined as the highest dose with no > grade 1 toxicity according to Common Toxicity Criteria (CTC).
  The dose-limiting toxicity (DLT) is defined as the dose, which leads with a 30% chance of toxicity to CTC Grade 2 or higher and / or leads to corrected QT interval (QTc)≥480ms and/or increase of QTc >= 50ms compared to baseline

SECONDARY OUTCOMES:
Incidence of treatment - Emergent Adverse Events (Safety) | during dose escalation and during 4 weeks treatment with MTD every week
  The analysis of safety assessments will include the following data collected for each subject:
  - Adverse Events (AEs) in the context of Drug Exposure (days)
Quantification of Vorinostat concentration in blood - pharmacokinetics | d21 by 4 weeks treatment with MTD
  Blood and plasma area under the concentration time curve of Vorinostat from time zero to 8 hours postdose.
  The pharmacokinetic study will investigate the correlation between dose administered and concentration of Vorinostat in blood.
association of alterations in the genome-wide transcriptome profile with the dose administered, toxicity and treatment response - pharmacodynamics | d21 by 4 weeks treatment with MTD
  The genome-wide transcriptome profile will be determined as a pharmacodynamic surrogate parameter. Alterations between baseline and after dose administered will be compared. The pharmacodynamic study will investigate the correlation between dose administered, alterations in the genome-wide transcriptome profile as well as treatment responses (memory performance) and toxicities.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - German Center for Neurodegenerative Diseases, Bonn
  - University Medical Center Göttingen, Department of Psychiatry and Psychotherapy, Göttingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia AA, Koperniku A, Ferreira JCB, Mochly-Rosen D. Treatment strategies for glucose-6-phosphate dehydrogenase deficiency: past and future perspectives. Trends Pharmacol Sci. 2021 Oct;42(10):829-844. doi: 10.1016/j.tips.2021.07.002. Epub 2021 Aug 10. PMID 34389161